CLINICAL TRIAL: NCT01083121
Title: Post-Marketing Surveillance of Humira Injection in Korean Patients Under the "New-Drug Re-examination"
Brief Title: Surveillance of Humira Injection in Korean Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-053
Record Dates: First submitted 2010-02-24; First posted 2010-03-09 (Estimated); Results first posted 2013-08-20 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Crohn's Disease; Psoriasis
Keywords: Postmarketing Drug Surveillance
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Crohn Disease; Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: Participants who were prescribed with adalimumab per approved prescribing information of adalimumab in Korea.

SUMMARY:
Patients who take Humira as prescribed by physicians as per Korean label will be enrolled and observed in normal medical practice setting for not less than 3 months following first dose of Humira. Information on demographics, diagnosis and medical history, results of tuberculosis skin test, results of chest X-ray, Humira treatment information, concomitant medication, physician's global assessment for effectiveness, disease activity assessment for rheumatoid arthritis, disease activity assessment for Crohn's Disease, disease activity assessment for Psoriasis and adverse events will be recorded on case report forms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19 years and above) with one of the following indications:

  * Moderately to severely active rheumatoid arthritis or
  * active and progressive psoriatic arthritis when the response to previous disease-modifying anti-rheumatic drug therapy has been inadequate or
  * severe active ankylosing spondylitis who have had an inadequate response to conventional therapy or
  * severely active Crohn's disease who have had no response, intolerance or contraindication to corticosteroid therapy or immunosuppressants or
  * moderately to severely active psoriasis patients who have had no response, have intolerance or have contraindication to systemic therapies including cyclosporine, methotrexate or photochemotherapy (PUVA).
* Patients who give verbal or written authorization to use their personal and health data.

Exclusion Criteria:

- Patients with known hypersensitivity to adalimumab or any of its excipients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics, general hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1779 (Actual)
Dates: Start 2007-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Chee, MD, Study Director — AbbVie Ltd.
Locations (77):
- South Korea (77):
  - Site Reference ID/Investigator# 29724, Ansan
  - Site Reference ID/Investigator# 53586, Ansan
  - Site Reference ID/Investigator# 29729, Bucheon-si
  - Site Reference ID/Investigator# 29009, Bucheon-si
  - Site Reference ID/Investigator# 29726, Busan
  - Site Reference ID/Investigator# 29733, Busan
  - Site Reference ID/Investigator# 28582, Busan
  - Site Reference ID/Investigator# 5633, Busan
  - Site Reference ID/Investigator# 28608, Cheonan
  - Site Reference ID/Investigator# 28996, Cheonan
  - Site Reference ID/Investigator# 29735, Daegu
  - Site Reference ID/Investigator# 59287, Daegu
  - Site Reference ID/Investigator# 29278, Daegu
  - Site Reference ID/Investigator# 29279, Daegu
  - Site Reference ID/Investigator# 29007, Daejeon
  - Site Reference ID/Investigator# 29727, Daejeon
  - Site Reference ID/Investigator# 29745, Daejeon
  - Site Reference ID/Investigator# 48624, Daejeon
  - Site Reference ID/Investigator# 29075, Goyang
  - Site Reference ID/Investigator# 29042, Guri-si
  - Site Reference ID/Investigator# 59285, Guri-si
  - Site Reference ID/Investigator# 29731, Gwangju
  - Site Reference ID/Investigator# 81693, Gwangju
  - Site Reference ID/Investigator# 29732, Gwangju
  - Site Reference ID/Investigator# 29737, Gwangju
  - Site Reference ID/Investigator# 29742, Gwangju
  - Site Reference ID/Investigator# 28611, Gyeongju
  - Site Reference ID/Investigator# 29103, Iksan
  - Site Reference ID/Investigator# 29010, Incheon
  - Site Reference ID/Investigator# 28589, Jeju City
  - Site Reference ID/Investigator# 29080, Jeju City
  - Site Reference ID/Investigator# 29743, Jeollabuk-do
  - Site Reference ID/Investigator# 29082, Jeonju
  - Site Reference ID/Investigator# 29740, Jinju
  - Site Reference ID/Investigator# 29172, Masan
  - Site Reference ID/Investigator# 29436, Metropolitan City Daejon
  - Site Reference ID/Investigator# 28970, Pohang
  - Site Reference ID/Investigator# 29723, Seongnam
  - Site Reference ID/Investigator# 29722, Seongnam
  - Site Reference ID/Investigator# 29738, Seoul
  - Site Reference ID/Investigator# 53584, Seoul
  - Site Reference ID/Investigator# 59283, Seoul
  - Site Reference ID/Investigator# 29452, Seoul
  - Site Reference ID/Investigator# 29453, Seoul
  - Site Reference ID/Investigator# 53583, Seoul
  - Site Reference ID/Investigator# 29728, Seoul
  - Site Reference ID/Investigator# 29734, Seoul
  - Site Reference ID/Investigator# 29721, Seoul
  - Site Reference ID/Investigator# 29029, Seoul
  - Site Reference ID/Investigator# 29736, Seoul
  - Site Reference ID/Investigator# 59282, Seoul
  - Site Reference ID/Investigator# 29741, Seoul
  - Site Reference ID/Investigator# 29165, Seoul
  - Site Reference ID/Investigator# 29166, Seoul
  - Site Reference ID/Investigator# 29011, Seoul
  - Site Reference ID/Investigator# 48623, Seoul
  - Site Reference ID/Investigator# 63322, Seoul
  - Site Reference ID/Investigator# 29748, Seoul
  - Site Reference ID/Investigator# 53582, Seoul
  - Site Reference ID/Investigator# 29076, Seoul
  - Site Reference ID/Investigator# 29034, Seoul
  - Site Reference ID/Investigator# 29434, Seoul
  - Site Reference ID/Investigator# 29435, Seoul
  - Site Reference ID/Investigator# 29744, Seoul
  - Site Reference ID/Investigator# 29041, Seoul
  - Site Reference ID/Investigator# 29012, Seoul
  - Site Reference ID/Investigator# 66654, Seoul
  - Site Reference ID/Investigator# 59284, Seoul
  - Site Reference ID/Investigator# 29035, Seoul
  - Site Reference ID/Investigator# 59286, Seoul
  - Site Reference ID/Investigator# 53588, Suwon
  - Site Reference ID/Investigator# 29746, Suwon
  - Site Reference ID/Investigator# 29739, Taegu
  - Site Reference ID/Investigator# 29085, Uljeongbu
  - Site Reference ID/Investigator# 28610, Ulsan
  - Site Reference ID/Investigator# 29725, Ulsan
  - Site Reference ID/Investigator# 29730, Wŏnju

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab
Started | 1779 (Participants who were enrolled in the study)
Completed | 1698 (Participants included in the analysis)
Not Completed | 81
Not completed — Use of Humira outside the approved label | 81

BASELINE CHARACTERISTICS:
Population: Safety analysis population
Arm/Group | Adalimumab
Number analyzed (Participants) | 1698
Age Continuous [Mean (Standard Deviation); unit: years] | 41.80 (13.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 729
  Male | 969
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 1,698
Indication [Number; unit: participants]
  Rheumatoid arthritis | 652
  Psoriatic arthritis | 47
  Ankylosing spondylitis | 925
  Crohn's disease | 73
  Psoriasis | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. An Adverse Drug Reaction (ADR) is any noxious and undesired reaction related to an experimental drug or experiment. A serious AE (SAE) is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome. AEs were rated for severity as either Mild: transient and easily tolerated; Moderate: causes discomfort and interrupts usual activities; or Severe: causes considerable interference with usual activities, may be incapacitating or life-threatening. AEs related to adalimumab were assessed as being either probably or possibly related by the investigator. An Unexpected ADR is an ADR for which the nature or gravity is not consistent with the applicable product information.
Time Frame: From Baseline until up to 70 days after the 3 month study period (total of 160 days).
Population: Safety analysis population
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 1698
participants
  Any adverse event | 171
  Any adverse drug reaction | 116
  Serious adverse events | 47
  Mild adverse event | 115
  Moderate adverse event | 58
  Severe adverse event | 7
  Discontinued adalimumab due to adverse event | 30
  Adverse events related to adalimumab | 120
  Unexpected adverse drug reaction | 21

2. Secondary Outcome: Physician's Global Assessment for Effectiveness
Description: The investigator's overall assessment for effectiveness was recorded as 'Improved', 'No change', 'Aggravated,' or 'Not assessable'.
Time Frame: After 3-month treatment
Population: Effectiveness evaluation was performed in 1,471 participants who received adalimumab for at least 3 months and in whom investigator's assessment at 3 months was available. No participants were available in the Psoriasis group for effectiveness evaluation.
Measure: Number; unit: participants
Groups:
- Rheumatoid Arthritis: Participants with moderately to severely active rheumatoid arthritis who were prescribed with adalimumab per approved prescribing information of adalimumab in Korea.
- Psoriatic Arthritis: Participants with active and progressive psoriatic arthritis who were prescribed with adalimumab per approved prescribing information of adalimumab in Korea.
- Ankylosing Spondylitis: Participants with severe active ankylosing spondylitis who were prescribed with adalimumab per approved prescribing information of adalimumab in Korea.
- Crohn's Disease: Participants with severely active Crohn's disease who were prescribed with adalimumab per approved prescribing information of adalimumab in Korea.
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis | Crohn's Disease
Number analyzed (Participants) | 541 | 40 | 834 | 56
participants
  Improved | 478 | 37 | 790 | 50
  No change | 52 | 2 | 41 | 6
  Aggravated | 11 | 1 | 3 | 0
  Not assessable | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For up to 70 days after the 3 month study period (total of 160 days).
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 47/1698
Other Adverse Events (participants affected / at risk) | 0/1698
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=1698)
Pyelonephritis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Peritoneal tuberculosis (Infections and infestations) | 2
Tuberculosis (Infections and infestations) | 2
Renal tuberculosis (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Malaria (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Intestinal infarction (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Pain (General disorders) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Knee operation (Surgical and medical procedures) | 1
Small intestinal resection (Surgical and medical procedures) | 1
Blood creatinine increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Allergy to sting (Immune system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.